CLINICAL TRIAL: NCT06061211
Title: Treadmill Training with TENS Impact on Walking Distance, Pain and Peak Velocity in Patients with Peripheral Arterial Disease
Brief Title: Treadmill with TENS on Functional Capacity &muscle Oxygenation in PAD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Kamal Abdelazim Hussein Elhashash, Assisstant lecturer of physical therapy for cardiovascular, respiratory and geriatrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NO:P.T.REC/012/004528
Record Dates: First submitted 2023-09-03; First posted 2023-09-29 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Intermittent Claudication; treadmill; TENS; Muscle oxygen saturation; Peak Systolic Velocity
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treadmill with TENS training (Experimental): SIDEA-Germany treadmill & MH8001 Portable tens Treadmill walking initially will begin exercising at 2 mph (3.2 km/h) at a 0% grade. They will walk until their claudication pain and determine site of pain then we will apply TENS on pain site and starting frequency at 2 HZ, then will increase inclination of treadmill gradually together with increasing frequancy of TENS up to 120 HZ if patient will report any feeling of pain, pain became moderately severe (4 of 5 on the claudication scale), throughout 45-minute exercise session. When a participant will be able to walk for 8 minutes at the initial workload without having to stop because of moderately severe claudication, the treadmill grade will be increased by increments of 0.5% until an 8-10% grade will be achieved. Subsequently, exercise intensity will be increased during training sessions by increasing the treadmill speed by increments of 0.1-0.2 mph (0.2-0.3 km/h) as tolerated
  Interventions: Other: TREADMILL(SIDEA-Germany treadmill ) with TENS
- Treadmill training (Other): Over the past 30 years, treadmill-based SET programs have been shown to be consistently beneficial in improving walking ability as assessed by graded treadmill testing and to be effective in patients with PAD both with and without classic symptoms of claudication. Treadmill-based exercise therapy for patients with PAD consists of intermittent bouts of walking exercise to moderate to moderately severe discomfort (4 of 5 on the claudication scale) followed by short periods of rest until symptoms resolve. These exercise/rest bouts are repeated over a 30- to 45-minute exercise session. Exercise capability is most commonly measured as COT/COD and PWT/PWD.
  Interventions: Other: TREADMILL(SIDEA-Germany treadmill ) with TENS

INTERVENTIONS:
Other: TREADMILL(SIDEA-Germany treadmill ) with TENS — TENS:
  MH8001 Portable tens 45 min. three times/ week 2-120 HZ 200ms
  treadmill: SIDEA-Germany treadmill three times/week, 45min, moderate intensity according to claudication pain scale 2MPH(3.5KM/h) 0% grade then increase by 2% every 2min.

SUMMARY:
Fifty patients from both sexes with PAD, stage II fontaine will participate in this study. Their ages will be from 40-75 years old. They will be selected from kasr el ainy (faculty of medicine), Cairo University, Giza, Egypt. The patients will be randomly assigned into two equal groups:

Group (A): 25 patients will receive transcutaneous electrical nerve stimulation (TENS) for 45 minutes per session applied on calf muscle, combined with treadmill three days per week for twelve weeks in addition to the routine medical treatment.

Group (B): 25 patients will receive treadmill training for 45 minutes per session, three days per week for twelve weeks in addition to the routine medical treatment

DETAILED DESCRIPTION:
Procedures of the study:

a) Evaluating procedures: It will be performed before treatment and 12 weeks after treatment program.

History and physical examination:

Complete history taking will be conducted to collect data about patient's general condition, current medication, measuring blood pressure, heart rate and physical activity.

Anthropometric measurement:

Weight and height will be measured for each patient in both groups. BMI will be calculated as follows: BMI (kg/m2) = Weight (kg) / Height (m2).

(FULLMEDI, FM-S120, China)

Ankle-brachial pressure index (ABI) :

is a useful screening test for detecting PAD. ABI value less than 0.9 is generally thought to have arterial stenosis or obstruction in lower limbs. However, Accurate ABI values may not be obtained and pseudo-normalize in cases of high arterial calcification or incompressible arteries, The resting ABI for each leg will be calculated by dividing the highest ankle systolic blood pressure (posterior tibial or dorsalis pedis) by the highest brachial systolic blood pressure; all resting pressures will be measured using a Doppler device at least 5 minutes after the patient will be rested quietly in the supine position.

ABPI Interpretation >1.3 Consider presence of calcification 1.0-1.3 Likely normal 0.9-1.0 Possible mild disease, borderline PAD 0.5-0.9 Claudication 0.3-0.5 Severe occlusive disease <0.3 Critical limb ischemia

Doppler ultrasonography: (a General Electric Logic P6 machine equipped with a linear probe with 7.5-12 MHz frequency and a curvilinear probe with 2.5-7.5 MHz frequency) It will be used to detect moving reflectors. Ultrasonography has the advantage of non-invasively measuring blood flow velocity in a quick and continuous manner based on the velocity of sound. Moreover, it enables examination of the state of the blood vessels from the vessel cross-section.

Duplex scanning will be performed by an experienced operator. APSV is the mean of the peak systolic velocities of the anterior and posterior tibial arteries (PTAs) measured at the ankle level. A 5-MHz convex probe will be used for the aorta and iliac arteries, and a 5- to 12-MHz linear transducer will be used for infrainguinal arteries. The Doppler angle of insonation will be adjusted to 60 μ. All patients will be rested 1 h before scanning and will be examined in supine position. Recordings will be made with the room temperature adjusted to 22°C. Peak systolic velocities of the distal PTA at or below the malleolar level and the distal anterior tibial artery (ATA) just above the ankle joint level will be recorded. Peak systolic velocities will be averaged over three cardiac cycles. If focal stenotic lesion will be detected in one of the distal tibial arteries, velocity measurements will be taken distal to the stenosis. No alterations will be made to the patient's medications before scanning .

Skeletal muscle oxygen saturation (SmO2) (Moxy, Fortiori Design LLC, Minnesota) Growing evidence suggests that changes in the microvasculature and skeletal muscle metabolism of oxygen in the leg contribute to claudication in PAD .Near-infrared spectroscopy (NIRS) will measure skeletal muscle oxygen saturation (SmO2) noninvasively. Smo2 will be measured from the capillaries in the muscle and is indicative of tissue oxygenation. Several studies suggest that the fall in leg Smo2 during walking is greater and occurs faster in PAD patients compared with healthy people.

A measure of muscle oxygen saturation, at the medial gastrocnemius in both legs of every participant. The Moxy uses continuous-wave spectroscopy which uses light of constant intensity that travels through the tissue and is collected by the receiver a certain distance away from the light source, SmO2 level measures with more sensitivity to the muscle layer and less sensitivity to the fat layer. Moxy in particular has source and receiver distance of 12 and 25 mm, which means it can penetrate into the tissue down to 12.5 mm. To make sure the NIRS device was collecting reliable SmO2 levels.

Treadmill exercise testing:

A graded treadmill test was used to assess walking capacity. Patients performed a progressive graded cardiopulmonary treadmill test until maximal claudication pain. The test started at 2 mph with 0% grade and the workload was increased 2% every 2 minutes. All patients were informed of the test protocol before being submitted to it. The results of the tests will be expressed in units of distance that will be walked up to the claudication pain (initial claudication distance) and the maximally tolerated claudication pain (maximal claudication distance). To exclude the training effect of treadmill, testing will be performed only once before and once after the procedure. However, before testing, patients will informed by the detailed instructions.

Maximal Treadmill Walking Time:

Change in maximal treadmill walking time will be measured at baseline, 12-week follow-up, using the Gardner-Skinner protocol.The treadmill test will begin at a speed of 2.0 miles per hour with 0 grade. Grade will increase by 2% every 2 minutes until the participant will not continue walking. When participants will be unable to walk at 2.0 miles per hour, the treadmill speed will start at 0.5 miles per hour and will increase by 0.5 miles per hour every 2 minutes until the treadmill will reach 2.0 miles per hour, after which the grade will be increased by 2% every 2 minutes. For maximum treadmill walking time, a small minimum clinically important difference will be defined as 38 seconds, and a large minimum clinically important difference will be defined as 152 seconds.

The Walking Estimated Limitation Calculated by History (WELCH) questionnaire: Each patient will be provided a pen and reading glasses (if needed) and will receive oral instructions on completing the questionnaire on arrival at the laboratory. Each patient will self-completed the questionnaires in the waiting room of the laboratory before the walking test will be performed. The questionnaire includes date of the visit, history and ongoing treatments, name and surname, age, sex, body weight, stature, active smoking, and the WELCH. The WELCH is a four item questionnaire that can be self-administered. The original questionnaire was developed in French but is currently available in various languages. In brief, the first three items refer to the maximum time that can be sustained when walking at different walking speeds. Answers to each item include proposals ranging from impossible (0 points) to 3 h or more (7 points). The fourth and last item requires the patient to estimate his/her usual walking speed as compared with that of his/her siblings or of people of comparable age. Possible answers will range from "much slower" (coefficient = 1) to "faster" (coefficient = 5). The WELCH score will be calculated as follows. One will be subtracted from the sum of the points of the three first items. The result of this subtraction will be multiplied by the coefficient of item four. the final score will range from 0 (severe disability) to 100 (ability to walk faster than other people for at least 3 h). Note that patients will never reminded of their answers to the previously completed WELCH questionnaires or their previous walking distance on the treadmill.

Short-physical performance battery:

The short physical performance battery is a group of measures that will combine the results of gait speed, chair stand, and balance tests:

* The standing balance test will require patients to maintain for 10 s in each stance, with their feet will be placed side by side, semi-tandem, and in tandem. For each stand, first we will demonstrate the task. Next, will support patients to maintain balance while they will position their feet, ask if they will be ready, release the support, and will begin timing. The timer will stop when participants move their feet or grasp the interviewer for support, or when 10 s will elapse. Scores will range from 0 to 4 (maximum performance).
* The chair stand test patients will stand up from a chair with their arms across their chest, five times, as quickly as possible. The patients will be timed from the initial sitting position to the final standing position at the end of the fifth stand. The time will be measured in seconds will be the outcome. Scores will range from 0 to 4 (maximum performance).
* The usual and fast gait speed of the patients over 4 m will be recorded using a stopwatch (within 0.1 s). To access their usual gait speed, patients will be instructed to "walk to the other end of the course at your usual speed, just as if you will walk down the street to go to the store." To access their fast gait speed, patients will be required to walk as fast as they can until the end of the course. Each patient will perform two timed attempts for both usual and fast gait speeds. The fastest walk of each pair (usual and fast) will be retained for analysis.

Scores will range from 0 to 4 (maximum performance). The total score from the physical performance battery will be calculated from the performance in the three tests, will range from 0 to 12, with 0 as worst function and 12 as best function.

Health-related quality of life (HRQOL) in patients with peripheral artery disease (PAD) (QOLPAD):

The QOLPAD is a short and feasible disease-specific instrument that can be used to evaluate HRQOL in patients with PAD in clinical routine or research. The new QOLPAD showed good psychometric properties, including high internal consistency at both measurement time points and convergent validity regarding the HRQOL of generic and disease-specific instruments. The one-page QOLPAD consisted of 12 questions with a five-step response scale. the QOLPAD evaluates current HRQOL impairment. Assessing the QOLPAD both before and after treatment allows detection of the improvement that can be assigned to the treatment.

B) Therapeutic equipment:

Transcutaneous electrical nerve stimulation TENS:

TENS machine will be fitted to the participant before walking on treadmill and continue for 45 minutes, it will be at low frequency at the beginning then if patients feel pain, then increasing frequency. A segmental electrode application will be used using self-adhesive carbon rubber electrodes measuring 5 * 5 cm. The 2 electrodes will be attached to the TENS unit via the manufacturer leads. The area of pain will be reported by the participant during the familiarization session will determine the electrode placement sites. The placement sites will be at least 2 cm apart. Electrodes will be commonly placed with 1 proximal and 1 distal to the gastrocnemius muscle belly. The HF-TENS stimulation parameters will be calibrated to 120 Hz, pulse width of 200 microseconds, and patient-will determine intensity of ''strong but comfortable.'' The LF-TENS stimulation will be set at 2 Hz, pulse width of 200 microseconds, and patient- will determine intensity of ''strong but comfortable and slight muscle twitch.

Treadmill:

Treadmill walking initially will begin exercising at 2 mph (3.2 km/h) at a 0% grade. They will walk until their claudication pain and determine site of pain then we will apply TENS on pain site and starting frequency at 2 HZ, then will increase inclination of treadmill gradually together with increasing frequancy of TENS up to 120 HZ if patient will report any feeling of pain, pain became moderately severe (4 of 5 on the claudication scale), throughout 45-minute exercise session. When a participant will be able to walk for 8 minutes at the initial workload without having to stop because of moderately severe claudication, the treadmill grade will be increased by increments of 0.5% until an 8-10% grade will be achieved. Subsequently, exercise intensity will be increased during training sessions by increasing the treadmill speed by increments of 0.1-0.2 mph (0.2-0.3 km/h) as tolerated.

ELIGIBILITY:
Inclusion Criteria:

* • Fifty patients who had intermittent claudication secondary to PAD

  * Ambulation during a graded treadmill test limited by leg pain consistent with intermittent claudication (stage II of the Fontaine classification of PAD)
  * Ankle-brachial index (ABI) of 0.90 or lower at rest or 0.73 or lower after exercise
  * Their age will be ranged from 40-75 years old
  * Body mass index (BMI) from 18.5 to 40 kg/m2
  * they are able to take part in an outpatient rehabilitation program
  * they are clinically stable
  * they are sedentary activity level according to Global Physical Activity Questionnaire (GPAQ).
  * smokers

Exclusion Criteria:

* • Absence of PAD

  * Inability to obtain an ABI measure because of non compressible vessels
  * Asymptomatic PAD determined from the medical history and verified during the graded treadmill test
  * Use of cilostazol and pentoxifylline initiated within 3 months before the investigation
  * Exercise tolerance limited by factors other than leg pain
  * Active cancer, renal disease, or liver disease
  * The presence of a contraindication to the use of TENS, such as a pacemaker or skin lesion.
  * walking disorders related to orthopedic or neuromuscular disease
  * myopathy
  * associated progressive disease causing deterioration in general health
  * implanted pacemaker or defibrillator
  * uncontrolled diabetes

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Doppler ultrasonography | 12 weeks( three months)
  Doppler ultrasonography: (a General Electric Logic P6 machine equipped with a linear probe with 7.5-12 MHz frequency and a curvilinear probe with 2.5-7.5 MHz frequency ) Duplex ultrasound (DUS) is an integral component of diagnostic testing for the evaluation and management of arterial disease. this technology, which combines the acquisition of blood flow (pulsed Doppler spectral analysis) and anatomic (B-mode and color Doppler imaging) ultrasonography has the advantage of non-invasively measuring blood flow velocity in a quick and continuous manner based on the velocity of sound. DUS rapidly expanded into peripheral arterial, visceral arterial, and peripheral venous applications, Duplex scanning will be performed by an experienced operator.
  APSV is the mean of the peak systolic velocities of the anterior and posterior tibial arteries (PTAs) measured at the ankle level.

SECONDARY OUTCOMES:
Treadmill exercise testing | 12 weeks( three months)
  to measure walking distance
Maximal Treadmill Walking Time | 12 weeks( three months)
  to measure walking time
Ankle brachial pressure index (ABI) | 12 weeks( three months)
  is a useful screening test for detecting PAD
The Walking Estimated Limitation Calculated by History (WELCH) questionnaire: to estimate walking capacity | 12 weeks( three months)
  Assess walking limitation in PAD
Quality of Life questionnaire for patients with peripheral artery disease, QOLPAD | 12 weeks( three months)
  evaluate HRQoL in patients with PAD
Skeletal muscle oxygen saturation (SmO2) | 12 weeks( three months)
  Near-infrared spectroscopy (NIRS) will measure skeletal muscle oxygen saturation (SmO2) noninvasively.
  A measure of muscle oxygen saturation, at the medial gastrocnemius in both legs of every participant. The Moxy uses continuous-wave spectroscopy which uses light of constant intensity that travels through the tissue and is collected by the receiver a certain distance away from the light source, SmO2 level measures with more sensitivity to the muscle layer and less sensitivity to the fat layer. Moxy in particular has source and receiver distance of 12 and 25 mm, which means it can penetrate into the tissue down to 12.5 mm. To make sure the NIRS device was collecting reliable SmO2 levels
Short-physical performance battery | 12 weeks( three months)
  The short physical performance battery is a group of measures that will combine the results of gait speed, chair stand, and balance tests: assess functional capacity
  • The usual and fast gait speed of the patients over 4 m will be recorded using a stopwatch (within 0.1 s). To access their usual gait speed, patients will be instructed to "walk to the other end of the course at your usual speed, just as if you will walk down the street to go to the store." To access their fast gait speed, patients will be required to walk as fast as they can until the end of the course. Each patient will performe two timed attempts for both usual and fast gait speeds. The fastest walk of each pair (usual and fast) will be retained for analysis.
  Scores will range from 0 to 4 (maximum performance). The total score from the physical performance battery will be calculated from the performance in the three tests, will range from 0 to 12, with 0 as worst function and 12 as best function

CONTACTS AND LOCATIONS:
Overall Officials: Hadeer K Elhashash, AL, Principal Investigator — faculty of physical therapy; Azza A ABDELHADY, Professor, Study Chair — faculty of physical therapy; Marwa M Elsayed, lecturer, Study Director — faculty of physical therapy; AHMED A SHAKER, AP, Study Director — Faculty of medecine; ASMAA H HABIB, Lecturer, Study Director — Faculty of medecine
Locations (1):
- Faculty of physical therapy, cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abaraogu UO, Dall PM, Brittenden J, Stuart W, Tew GA, Godwin J, Seenan CA. Efficacy and Feasibility of Pain management and Patient Education for Physical Activity in Intermittent claudication (PrEPAID): protocol for a randomised controlled trial. Trials. 2019 Apr 16;20(1):222. doi: 10.1186/s13063-019-3307-6. PMID 30992033
- [Background] Aboyans V, Ricco JB, Bartelink MEL, Bjorck M, Brodmann M, Cohnert T, Collet JP, Czerny M, De Carlo M, Debus S, Espinola-Klein C, Kahan T, Kownator S, Mazzolai L, Naylor AR, Roffi M, Rother J, Sprynger M, Tendera M, Tepe G, Venermo M, Vlachopoulos C, Desormais I; ESC Scientific Document Group. 2017 ESC Guidelines on the Diagnosis and Treatment of Peripheral Arterial Diseases, in collaboration with the European Society for Vascular Surgery (ESVS): Document covering atherosclerotic disease of extracranial carotid and vertebral, mesenteric, renal, upper and lower extremity arteriesEndorsed by: the European Stroke Organization (ESO)The Task Force for the Diagnosis and Treatment of Peripheral Arterial Diseases of the European Society of Cardiology (ESC) and of the European Society for Vascular Surgery (ESVS). Eur Heart J. 2018 Mar 1;39(9):763-816. doi: 10.1093/eurheartj/ehx095. No abstract available. PMID 28886620
- [Background] Aday AW, Lawler PR, Cook NR, Ridker PM, Mora S, Pradhan AD. Lipoprotein Particle Profiles, Standard Lipids, and Peripheral Artery Disease Incidence. Circulation. 2018 Nov 20;138(21):2330-2341. doi: 10.1161/CIRCULATIONAHA.118.035432. PMID 30021845
- [Background] Arman EB, Augustin M, Mohr N, Debus SE, Breuer P, Blome C. Development and validation of a disease-specific quality of life questionnaire for patients with peripheral artery disease (QOLPAD). J Patient Rep Outcomes. 2022 May 27;6(1):54. doi: 10.1186/s41687-022-00451-0. PMID 35622190